CLINICAL TRIAL: NCT00104819
Title: Phase II Trial of FavId™ (Patient-Specific Idiotype/KLH) and GM-CSF in Subjects Who Demonstrated Progressive Disease and Did Not Receive FavId on Study FavId-06
Brief Title: Vaccine Therapy and GM-CSF in Treating Patients With Progressive Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn as company has shut down and filed for bankruptcy
Sponsor: Favrille (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: FAV-ID-09; CDR0000415573 (Registry Identifier: PDQ (Physician Data Query)); CWRU-FVID-2404; CWRU-100415; CASE-2404; FAV-WIRB-20041124
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-08

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — sargramostim

INTERVENTIONS:
Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines made from a person's cancer cells may make the body build an effective immune response to kill cancer cells. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood and may stimulate the immune system in different ways and stop cancer cells from growing.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with GM-CSF works in treating patients with progressive B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Provide treatment with autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId)™ and sargramostim (GM-CSF) to patients with progressive grade 1, 2, or 3 follicular B-cell non-Hodgkin's lymphoma who did not receive FavId™ while enrolled on protocol FAV-ID-06.

Secondary

* Determine the response rate and duration of response in patients treated with this regimen.
* Determine the response rate and response rate improvement after best response to prior salvage therapy in patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 groups according to timing of disease progression while enrolled on protocol FAV-ID-06 (disease progression after prior rituximab AND never randomized vs disease progression after randomization to placebo arm).

Patients receive autologous immunoglobulin idiotype-KLH vaccine subcutaneously (SC) on day 1. Patients also receive sargramostim (GM-CSF) SC on days 1-4. Treatment repeats monthly for 6 months in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may receive additional treatment as above every 2 months for 1 year (6 treatments) and every 3 months until disease progression.

After completion of study treatment, patients are followed for 30 days or until the start of subsequent treatment.

PROJECTED ACCRUAL: Approximately 238 patients (67 in group I and 171 in group II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular B-cell non-Hodgkin's lymphoma (NHL)

  * Grade 1, 2, or 3
* Progressive disease AND did not receive autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId™) while enrolled on protocol FAV-ID-06
* Meets 1 of the following criteria:

  * Received salvage therapy after completion of protocol FAV-ID-06

    * At least 4 weeks, but no more than 4 months, since prior salvage therapy
  * Did not receive salvage therapy after completion of protocol FAV-ID-06

    * At least 4 weeks, but no more than 4 months, since completion of prior treatment on protocol FAV-ID-06
* No history of CNS lymphoma OR meningeal lymphomatosis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No history of congestive heart failure

Pulmonary

* No history of compromised pulmonary function

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active bacterial, viral, or fungal infection
* No psychiatric disorder
* No other serious nonmalignant disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior allogeneic transplantation*
* No prior rituximab regimen* other than that administered on protocol FAV-ID-06 (rituximab 375 mg/m^2 IV weekly for 4 weeks)

Chemotherapy

* No prior purine analogues* (e.g., fludarabine or cladribine)

Endocrine therapy

* No prior or concurrent steroids (e.g., steroid doses in excess of daily replacement)

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Recovered from prior salvage therapy
* No prior or concurrent immunosuppressive therapy
* No prior investigational agents*
* No other concurrent antilymphoma therapy NOTE: *As salvage therapy administered between completion of protocol FAV-ID-06 and enrollment onto this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2004-09; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId)™ provided to patients who did not receive autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId)™ during participation on study Favld-06

SECONDARY OUTCOMES:
Response rate by modified Cheson Criteria
Duration of response by modified Cheson Criteria
Time to progression
Response rate improvement

CONTACTS AND LOCATIONS:
Overall Officials: John F. Bender, PharmD, Study Chair — Favrille
Locations (51):
- United States (51):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Sharp Memorial Hospital Cancer Center, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Rocky Mountain Cancer Centers - Denver Midtown, Denver, Colorado
  - Helen F. Graham Cancer Center at Christiana Hospital, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Center for Hematology-Oncology - Boca Raton, Boca Raton, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Kootenai Cancer Center - Coeur d'Alene, Coeur d'Alene, Idaho
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Kaiser Permanente Medical Office - Interstate Medical Office Central, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
  - Cancer Care Centers of South Texas - Medical Center, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin